CLINICAL TRIAL: NCT00534404
Title: iQuit Smoking: A Randomized Trial of Internet Access to Nicotine Patches
Brief Title: A Randomized Trial of Internet Access to Nicotine Patches
Acronym: iQS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Lawrence C. An, Associate Professor of Internal Medicine, Medical School, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 511; R01HL086684-01 (NIH)
Record Dates: First submitted 2007-09-21; First posted 2007-09-24 (Estimated); Results first posted 2015-02-03 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-01

CONDITIONS: Smoking Cessation; Tobacco Use Disorder
Keywords: Internet-Assisted Tobacco Treatments; Online Smoking Cessation Programs; Nicotine Patches; Telephone Counseling; Smoking Abstinence
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder | interventions — Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- NRT Patch, Phone Counseling, Internet (Experimental): As adjuncts to internet-assisted tobacco treatment (iQuit Smoking website), research participants in this arm will have access to free 8-week supply of nicotine patches, contingent upon participation in proactive telephone counseling. Patch therapy will begin with the 21 mg patch for 4 weeks, followed by 14 mg patch for 2 weeks, then 7 mg patch for 2 weeks.
  Interventions: Drug: Nicotine patches; Behavioral: Telephone counseling; Behavioral: iQuit Smoking website
- Nicotine Patches and Internet (Active Comparator): As adjuncts to internet-assisted tobacco treatment (iQuit Smoking website), research participants in this arm will have access to free 8-week supply of nicotine patches. Patch therapy will begin with the 21 mg patch for 4 weeks, followed by 14 mg patch for 2 weeks, then 7 mg patch for 2 weeks.
  Interventions: Drug: Nicotine patches; Behavioral: iQuit Smoking website
- Internet (Placebo Comparator): Research participants in this arm will have free access to internet-assisted tobacco treatment (iQuit Smoking website).
  Interventions: Behavioral: iQuit Smoking website

INTERVENTIONS:
Drug: Nicotine patches — Participants will wear nicotine patches.
  Other Names: Nicoderm CQ
  Arms: NRT Patch, Phone Counseling, Internet; Nicotine Patches and Internet
Behavioral: Telephone counseling — Participants receiving telephone counseling will receive five phone calls over a 2-month period to discuss their personal smoking cessation plan.
  Arms: NRT Patch, Phone Counseling, Internet
Behavioral: iQuit Smoking website — Participants will access the Project Quit (iQuit Smoking) website.

SUMMARY:
People who smoke cigarettes have an increased risk of developing emphysema, heart disease, and certain types of cancer. This study will evaluate the effectiveness of providing free nicotine patches from an online smoking cessation program, with and without telephone counseling, at improving quit rates in cigarette smokers.

DETAILED DESCRIPTION:
The objective of this project is to determine the efficacy and cost-effectiveness of providing access to free nicotine patches, with or without a required linkage to proactive telephone counseling, as adjuncts to internet-assisted tobacco treatment. Online cessation services will be provided by the Center for Health Communication Research at the University of Michigan.

This investigation has three specific aims and one exploratory aim:

* Specific Aim 1: To determine the efficacy of providing access to free nicotine patches as an addition to online smoking cessation services.
* Specific Aim 2: To determine the efficacy of providing access to free nicotine patches linked with proactive telephone counseling as an addition to online smoking cessation services.
* Specific Aim 3: To determine the cost-effectiveness of providing access to free nicotine patches, with or without linkage to proactive phone counseling, as additions to online cessation services.
* Exploratory Aim 1: To examine potential mediators and moderators of intervention effects. An examination of potential mediators will identify key psychological and behavioral processes (e.g. medication adherence, self-efficacy, etc.) that underlie how the interventions affect the process of quitting and offer guidance regarding key targets for future research. An examination of potential moderators (e.g. level of dependence, income, gender) will identify candidate subgroups for which the proposed interventions may be more effective and cost- effective.

Smokers searching online for help quitting (N=2,475) will be recruited and randomized to receive one of three treatments:

1. online smoking cessation services (i.e. web),
2. online cessation services plus access to free nicotine patches (i.e.web+patch),
3. online cessation services with access to free patches contingent upon participation in proactive telephone counseling (i.e. web+patch+phone).

The Center for Health Communications Research at the University of Michigan will serve as the smoking cessation website for this research project. Developed by Vic Strecher and colleagues, Project Quit is a web-based program designed to help individuals who would like to quit smoking in the next 30 days. The program is grounded in cognitive-behavioral methods of smoking cessation and relapse prevention. The web-based smoking cessation intervention features highly tailored email messages. Once enrolled in the project and the baseline assessment is completed, participants receive six tailored web sessions namely:

* Action plan (1 week before quit date);
* Barriers 1 (2 days before quit date);
* Supportive message (on quit date);
* Barriers 2 (2 days after quit date);
* Motivation (1 week after quit date);
* Testimonial (2 weeks after quit date).

Evaluations will occur at baseline and at 1-, 3-, and 9-months post-enrollment. The primary outcome measure will be self-reported 6-month prolonged abstinence measured at the 9-month evaluation.

This proposal addresses a critical need for evidence-based cessation treatments for smokers. At the completion of this project, it is our expectation that we will have identified an effective online intervention package (or packages) for dissemination of internet-assisted tobacco treatment.

This study will enroll people recruited via online sources. Participants will complete a baseline survey about their smoking habits and quit history. Participants will then be randomly assigned to one of the following three treatment groups:

* Group 1 participants will receive access to an online tailored stop smoking program.
* Group 2 participants will receive free access to nicotine patches and an online tailored stop smoking program.
* Group 3 participants will receive telephone counseling, free access to nicotine patches and an online tailored stop smoking program.

Participants receiving telephone counseling will receive 5 phone calls over a 2-month period to discuss their personal smoking cessation plan; they must complete the pre-quit and 7-10 day calls in order to receive the nicotine patches. At 1, 3, and 9 months post-enrollment, all participants will complete online surveys about their smoking cessation experience. Participants will be contacted by phone to complete the surveys if they do not complete them online.

ELIGIBILITY:
Inclusion Criteria:

* Currently smokes 10 or more cigarettes per day
* Does not use any tobacco products other than cigarettes
* Willing to set a quit date within 2 to 4 weeks following study entry
* Willing to use a nicotine patch
* Able to speak English
* Access to Internet, email, and telephone at work or home
* Resident of the United States
* Only one person per household is eligible to enroll

Exclusion Criteria:

* Medically unable to use the nicotine patch (e.g., pregnant, history of a heart attack)
* Currently uses nicotine replacement therapy (NRT) products
* Currently uses or plans to use Bupropion SR, Wellbutrin, or Zyban

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2485 (Actual)
Dates: Start 2011-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence C An, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Interested individuals completed a screening survey to determine eligibility. Following study consent, participants completed two emailed surveys over the next two days and a phone confirmation call before being randomized. These check-ins confirmed the participant had valid contact information and maintained their desire to quit smoking.
Period: Overall Study
Arm/Group | NRT Patch, Phone Counseling, Internet | Nicotine Patches and Internet | Internet
Started | 827 | 830 | 828
Completed at Least 1 Online Session | 781 | 813 | 658
Completed First NRT Order | 765 | 821 (Participants could order NRT without completing a web session) | 0 (NRT was not available for this arm)
Completed Second NRT Order | 640 | 789 | 0 (NRT not available for this arm.)
Completed at Least 1 Counseling Call | 813 | 0 (There was no counseling offered in this arm) | 0 (There was no counseling offered in this arm)
1-month Follow up Completed | 742 | 781 | 626
3-month Follow up Completed | 682 | 731 | 593
Completed | 647 | 687 | 586
Not Completed | 180 | 143 | 242
Not completed — Death | 0 | 0 | 2
Not completed — Withdrawal by Subject | 8 | 2 | 38
Not completed — Removed by study staff | 2 | 3 | 1
Not completed — Lost to Follow-up | 170 | 138 | 201

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NRT Patch, Phone Counseling, Internet | Nicotine Patches and Internet | Internet | Total
Number analyzed (Participants) | 827 | 830 | 828 | 2485
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 796 | 791 | 800 | 2387
  >=65 years | 31 | 39 | 28 | 98
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.27 (12.03) | 44.31 (12.00) | 44.20 (11.64) | 44.26 (11.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 562 | 581 | 578 | 1721
  Male | 265 | 249 | 250 | 764
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30 | 33 | 33 | 96
  Not Hispanic or Latino | 797 | 797 | 795 | 2389
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 5 | 6 | 16
  Asian | 7 | 8 | 6 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 3 | 5
  Black or African American | 56 | 56 | 64 | 176
  White | 714 | 725 | 712 | 2151
  More than one race | 32 | 23 | 24 | 79
  Unknown or Not Reported | 13 | 11 | 13 | 37
Region of Enrollment [Number; unit: participants]
  United States | 827 | 830 | 828 | 2485
Highest education level [Number; unit: participants]
  High school or less | 236 | 206 | 201 | 643
  Some college | 440 | 463 | 481 | 1384
  College graduate | 151 | 161 | 146 | 458

OUTCOME MEASURES:

1. Primary Outcome: Self-reported 6-month Prolonged Abstinence From Smoking
Description: Participants complete the final study survey 9 months following enrollment in the program. They are asked to report when they had last smoked a cigarette, even a puff. Participants who report that they have not smoked in the past 6 months are counted as abstinent for the purposes of our study analysis.
Time Frame: Measured at 9 Months post-randomization
Population: All currently enrolled participants were invited via email to complete an online follow-up survey. Participants who did not respond to the email received phone calls from study staff asking them to complete the survey online. Results to this outcome measure are from those subjects who completed the survey.
Measure: Number; unit: participants
Arm/Group | NRT Patch, Phone Counseling, Internet | Nicotine Patches and Internet | Internet
Number analyzed (Participants) | 647 | 687 | 586
participants | 252 | 194 | 109

2. Secondary Outcome: Self-reported 30-day Prolonged Abstinence at 9-month Follow up
Time Frame: 9 months post randomization
Measure: Number; unit: participants
Arm/Group | NRT Patch, Phone Counseling, Internet | Nicotine Patches and Internet | Internet
Number analyzed (Participants) | 647 | 687 | 586
participants | 310 | 268 | 176

3. Secondary Outcome: Self-reported 30-day Prolonged Abstinence at 3-month Follow up
Time Frame: 3-months post randomization
Measure: Number; unit: participants
Arm/Group | NRT Patch, Phone Counseling, Internet | Nicotine Patches and Internet | Internet
Number analyzed (Participants) | 682 | 731 | 593
participants | 379 | 299 | 138

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a 3-year period, from March 2011-March 2014
Arm/Group | NRT Patch, Phone Counseling, Internet | Nicotine Patches and Internet | Internet
Serious Adverse Events (participants affected / at risk) | 3/827 | 0/830 | 2/828
Other Adverse Events (participants affected / at risk) | 0/827 | 0/830 | 0/828
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NRT Patch, Phone Counseling, Internet (N=827) | Nicotine Patches and Internet (N=830) | Internet (N=828)
Death (General disorders) | 0 (0) | 0 (0) | 2 (2) — Reports of participants' deaths were received third person after the fact. These adverse events were classified by the Institutional Review Board as unrelated to study, unexpected.
Hospitalization (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes